CLINICAL TRIAL: NCT03218943
Title: Physiological Dead Space Measured by Volumetric Capnography, Is it Different Between the Biphasic Positive Airway Pressure Mode ( BiPAP ) and Airway Pressure Release Ventilation Mode ( APRV ) ? A Randomized Controlled Study.
Brief Title: Physiological Dead Space Measured by Volumetric Capnography in BiPAP and APRV .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Samir Awad Elkahwagy, Principal Investigator ,Dr. Ahmed Samir Elkahwagy, Kasr El Aini Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: N-44-2017
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Ventilation Therapy; Complications
Keywords: BiPAP; APRV; Physiological dead space; volumetric capnography; ARDS; impaired oxygenation; ICU; Mechanical ventilation
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: A randomized controlled study with cross-over design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APRV ventilation (Active Comparator): They will start on APRV mode with high pressure (Phi) 20 cmH2O , low pressure(Plo) 5 cmH2O with I:E ratio ( Phi phase: Plo phase ratio ) 4:1 for 3 hours Then, they will return to the initial settings ( PCV ) for 2 hours . then, they will be switched into BiPAP mode with high pressure (Phi) 20 cmH2O , low pressure(Plo) 5 cmH2O with I:E ratio ( Phi phase: Plo phase ratio ) 1:1 for 3 hours. Then left for ventilation according to the preference of the physician in charge.
  Interventions: Device: APRV ventilation mode
- BiPAP ventilation (Active Comparator): They will start on BiPAP mode with high pressure (Phi) 20 cmH2O , low pressure(Plo) 5 cmH2O with I:E ratio ( Phi phase: Plo phase ratio ) 1:1 for 3 hours. Then, they will return to the initial settings ( PCV ) for 2 hours . then, they will be switched into APRV mode with high pressure (Phi) 20 cmH2O , low pressure(Plo) 5 cmH2O with I:E ratio ( Phi phase: Plo phase ratio ) 4:1 for 3 hours. Then left for ventilation according to the preference of the physician in charge.
  Interventions: Device: BIPAP ventilation moood

INTERVENTIONS:
Device: APRV ventilation mode — They will start on APRV mode with high pressure (Phi) 20 cmH2O , low pressure(Plo) 5 cmH2O with I:E ratio ( Phi phase: Plo phase ratio ) 4:1 for 3 hours
  Arms: APRV ventilation
Device: BIPAP ventilation moood — start on BiPAP mode with high pressure (Phi) 20 cmH2O , low pressure(Plo) 5 cmH2O with I:E ratio ( Phi phase: Plo phase ratio ) 1:1 for 3 hours
  Arms: BiPAP ventilation

SUMMARY:
Background and Rationale :

Mechanical ventilation is an essential component of the care of patients with respiratory failure.Biphasic positive Airway Pressure (BiPAP) and Airway Pressure release ventilation (APRV) are relatively new modes of mechanical ventilation which can be used in treatment of patients with impaired oxygenation.The effect of using BiPAP and APRV modes on reducing the physiological dead space had not been previously investigated. The investigators hypothesize that using APRV mode will decrease physiological dead space more than BiPAP mode in the mechanically ventilated critically ill patients.

Objectives :

To assess the physiological dead space with each mode. To assess lung mechanics during the use of the two modes. To assess the effectiveness of ventilation during the use of the two modes.

Study population & Sample size :

Sixty adult patients more than 18 years old who are mechanically ventilated patients with P/F ratio less than 300. This sample size was calculated based on the assumption that APRV will decrease dead space by 20% with alpha error 0.05 and power 80%. The mean and Standard deviation of the volume of the dead space assessed in a previous study using BIPAP was 40

Study Design :

A randomized controlled non-blinded study with cross-over design. In the Trauma and surgical ICU at 185-Hospital (Kasr Alainy Hospitals).

Methods :

All mechanically ventilated patients in Trauma and surgical ICU at 185-Hospital (Kasr Alainy Hospitals) will start on pressure controlled ventilation mode (PCV) with inspiratory pressure achieving tidal volume 6-8 ml/kg for 2 hours then they will be randomized into one of the two study groups the BIPAP group or the APRV group .

Possible Risk (s) to study population :

By adjusting the ventilator parameters properly and continuous monitoring of the patients in the study, there will be no risk facing the patients.

Outcome parameter (s):

Primary outcome: Physiological dead space will be measured in the two groups after 30 minutes.

Secondary outcomes

* Physiological dead space after 3 hours.
* PO2/FiO2 ratio.
* Peak airway and Mean airway pressures.
* PCO2 and PH.
* Dynamic compliance.

DETAILED DESCRIPTION:
All mechanically ventilated patients in Trauma and surgical ICU at 185-Hospital (Kasr Alainy Hospitals) will start on pressure controlled ventilation mode (PCV) with inspiratory pressure achieving tidal volume 6-8 ml/kg for 2 hours then they will be randomized into : A-group (APRV group) & B-group (BiPAP group). which are described later in the 2 arms of the study.

Measurement tools :

The following data will be recorded :

* Demographic data ( Age , Sex , Weight and Height ).
* P/F ratio before inclusion.
* All patients then will be connected to Volumetric capnography which is included in the metabolic module on General Electric ventilator (Engstrom Carestation, GE Health care, USA). and physiological dead space will be recorded after 30 minutes and at the end of the 3 hours on each APRV & BiPAP modes .
* Peak air way pressure.
* Mean airway Pressure. They will be also recorded after
* Dynamic Compliance. 30 Minutes and at the end of the
* P/F ratio , PH and pCO2. 3 hours On APRV & BiPAP modes.
* Minute ventilation.
* Blood pressure , Heart rate and central venous pressure will be recorded before inclusion . then , they will be also recorded every 2 hours .

ELIGIBILITY:
Inclusion Criteria:

* Adults above 18 years old.
* Patients who are recently mechanically ventilated ( within 48 hours ).
* Patients with P/F ratio less than 300.

Exclusion Criteria:

* patients with COPD or pneumothorax.
* Patients with acute lung injury.
* patients with Emphysema and Emphysematous bullae .
* patients with broncho-pleural fistula.
* patients with severe hemodynamic instability (on IV Noradrenaline > 0.8 mic/kg/min).
* patients with cardiomyopathy , and those with stenotic valvular diseases.
* Patients with increased intracerebral pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-25 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Physiological dead space | after 30 min. on each mode ( APRV and BiPAP )
  percentage of vd/vt ( dead space volume/ Tidal volume ) which is measured by volumetric capnography included in the metabolic module on General Electric ventilator (Engstrom Carestation, GE Health care, USA).

SECONDARY OUTCOMES:
Physiological dead space. | after 3 hours on each mode ( APRV and BiPAP ).
  percentage of vd/vt ( dead space volume/ Tidal volume ) which is measured by volumetric capnography included in the metabolic module on General Electric ventilator (Engstrom Carestation, GE Health care, USA).
PO2/FiO2 ratio | after 30 min. and 3 hours on each mode ( APRV and BiPAP ).
  PO2 from ABG / FiO2 set on the ventilator
Peak airway pressure | after 30 min. and 3 hours on each mode ( APRV and BiPAP ).
  measured by the ventilator in cmH2O.
Mean airway pressure | after 30 min. and 3 hours on each mode ( APRV and BiPAP ).
  measured by the ventilator in cmH2O.
Dynamic compliance | after 30 min. and 3 hours on each mode ( APRV and BiPAP ).
  measured by the ventilator ml/cmH2O
PCO2 | after 30 min. and 3 hours on each mode ( APRV and BiPAP ).
  from ABG
pH | after 30 min. and 3 hours on each mode ( APRV and BiPAP ).
  from ABG

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkahwagy, Study Director — Department of Anesthesia , intensive care and pain management at kasr Alainy hospitals -faculty of medicine - Cairo Uni. - Egypt
Locations (1):
- Department of Anesthesia , intensive care and pain management -faculty of medicine Cairo Uni.- kasr Alainy Hospitals., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haitsma JJ, Lachmann RA, Lachmann B. Lung protective ventilation in ARDS: role of mediators, PEEP and surfactant. Monaldi Arch Chest Dis. 2003 Apr-Jun;59(2):108-18. PMID 14635498
- [Background] Hormann C, Baum M, Putensen C, Mutz NJ, Benzer H. Biphasic positive airway pressure (BIPAP)--a new mode of ventilatory support. Eur J Anaesthesiol. 1994 Jan;11(1):37-42. PMID 8143712
- [Background] Baum M, Benzer H, Putensen C, Koller W, Putz G. [Biphasic positive airway pressure (BIPAP)--a new form of augmented ventilation]. Anaesthesist. 1989 Sep;38(9):452-8. German. PMID 2686487
- [Background] Verscheure S, Massion PB, Verschuren F, Damas P, Magder S. Volumetric capnography: lessons from the past and current clinical applications. Crit Care. 2016 Jun 23;20(1):184. doi: 10.1186/s13054-016-1377-3. PMID 27334879
- [Background] Anderson CT, Breen PH. Carbon dioxide kinetics and capnography during critical care. Crit Care. 2000;4(4):207-15. doi: 10.1186/cc696. Epub 2000 Jul 12. PMID 11094503
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/14635498
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/8143712
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/2686487
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27334879
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/11094503